CLINICAL TRIAL: NCT06972901
Title: Evaluation of Therapeutic Strategy to Prevent Crohn's Disease Endoscopic poSToperatIve recurreNce Based on earlY Dosage of Faecal Calprotectin
Acronym: DESTINY II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOI 2022 BUISSON (DESTINY II); 2024-A02839-38 (Other: 2024-A02839-38)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease (CD); Ileocolic Resection; Post-endoscopic Operative Reccurence
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): Early dosage of fecal calprotectin at 3 months
  Interventions: Biological: Early faecal calprotectin dosage
- Standard arm (No Intervention): Standard dosage of fecal calprotectin at 6 months

INTERVENTIONS:
Biological: Early faecal calprotectin dosage — An early dosage of faecal calprotectin will be done for the active arm group.
  Arms: Active arm

SUMMARY:
Crohn's disease (CD) (> 200,000 patients in France) is a chronic inflammatory disease that can lead to progression of intestinal destruction and impaired quality of life. Despite the widespread use of biotherapies, intestinal resections remain frequent (50% of patients over time). Unfortunately, surgery is not curative since 75% of patients experienced post-endoscopic operative recurrence (POR) (i.e., recurrence of ulcerations) during the first year after surgery. Prevention of endoscopic POR (defined as a Rutgeerts index ≥ i2) is essential because endoscopic POR is highly predictive of clinical POR (i.e., recurrence of CD-related symptoms): > 40% and > 80% within 5 years for a Rutgeerts index ≥ i2 or ≥ i3, respectively. The recommended management is to start treatment after surgery to avoid endoscopic POR, and to perform a colonoscopy at 6 months (M6) with therapeutic escalation if endoscopic POR. Despite anti-TNF or ustekinumab treatment, the endoscopic POR rate remains high (30-40% at M6) leading to > 40% clinical POR despite therapeutic escalation (90 mg/4 weeks with ustekinumab) potentially due to late therapeutic escalation. Innovative strategies are therefore needed to prevent endoscopic POR, such as the use of fecal calprotectin, a non-invasive biomarker associated with endoscopic CD activity. We have previously demonstrated that its variation between surgery and M3 allows for a value at M3 predictive of endoscopic POR at M6. In this study, we hypothesize, for the first time, that a strategy integrating fecal calprotectin measurement at M3 with earlier therapeutic escalation (M3 vs M6) in case of abnormal value or kinetics could decrease the rate of endoscopic POR at M6.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter, two-arm, randomized, controlled clinical trial evaluating innovative versus standard care in patients with Crohn's disease. All eligible patients will be offered the study consecutively by the principal investigator or any other co-investigator declared on the study.

At the pre-inclusion visit (W-4 to W0 before inclusion), after verification of inclusion and non-inclusion criteria and obtaining consent, a laboratory assessment and an abdominal ultrasound (if participating in the DESTINY-echo ancillary study) will be prescribed (pre-biotherapy assessment, CRP) as well as a fecal calprotectin measurement.

After reverifying the inclusion and non-inclusion criteria, at the inclusion visit (W0), patients will be randomized between the two study arms (standard arm vs. active arm). Randomization will be stratified by center and number of risk factors. The results of this randomization will be shared with both the investigator and the patient.

The reference arm will be based on daily practice, i.e., regular monitoring (weeks 0 and 24) with fecal calprotectin testing at week 10, the results of which will be unknown for the duration of the study but may be disclosed upon patient exit, and with ustekinumab intensification at 6 months based on endoscopy results. In the active arm, in the event of an abnormal fecal calprotectin test result (> 100 μg/g at week 10 or a variation between week 0 and week 10 of > 50 μg/g), the investigator will be informed by electronic alert, and treatment intensification at week 12 will be required. Fecal calprotectin testing will be standardized and performed using the same test in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of CD according to ECCO guidelines
* Adult Crohn's disease (age ≥ 18 years)
* Having undergone ileal, colonic, or ileocolonic resection without residual macroscopic lesions
* With an anastomosis that can be reached by ileocolonoscopy
* With at least one of the following risk factors for endoscopic POR: active smoking, previous intestinal resection (before the current resection), length of resected small bowel > 30 cm, fistulizing phenotype (B3 according to the Montreal classification), exposure to at least two biotherapies before surgery
* No contraindication to ustekinumab treatment
* Patient capable of giving consent
* Patient covered by the French healthcare system

Exclusion Criteria:

* Permanent stoma
* Total colectomy
* Uncontrolled postoperative infectious complication
* Pregnant or breastfeeding women: a pregnancy test will be performed for women of childbearing age
* Refusal to participate in the study
* Persons deprived of their liberty by judicial or administrative decision
* Minors
* Vulnerable protected adults (under guardianship, curatorship, or legal protection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative endoscopic recurrence | 6 months post-operative
  Postoperative endoscopic recurrence at 6 months, defined by a Rutgeerts index ≥ i2.
  This primary endpoint will be defined by endoscopic procedure at 6 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Buisson, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (8):
- France (8):
  - CHU d'Amiens, Amiens
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Lille, Lille
  - HCL, Lyon
  - AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - Chu de Nice, Nice
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No